CLINICAL TRIAL: NCT01021124
Title: A Prospective Observational Study of Usefulness of a T Cell-based Assay for Latent Tuberculosis Infection in Hematopoietic Stem Cell Transplant Recipients
Brief Title: Latent Tuberculosis Infection in Bone Marrow Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assistant Professor, Asan Medical Center
Other Study IDs: 2009-0077
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Tuberculosis
Keywords: tuberculosis; bone marrow transplant; diagnosis
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- QFT (+) vs QFT (-)

SUMMARY:
The aim of this study is to estimate the usefulness of a T cell-based assay (i.e. Quantiferon-Gold In-Tube assay) for diagnosis of latent tuberculosis infection (LTBI) in bone marrow transplant recipients. For this purpose, the investigators enrolled bone marrow transplant recipients and observed the developement of tuberculosis after the transplantation.

DETAILED DESCRIPTION:
All adult bone marrow transplant recipients admitted to Asan Medical Center will be enrolled.

Quantiferon-Gold In-Tube assay will be performed.

Isoniazid prophylaxis will be given only to patients with clinical risk factors (i.e. recent contact with active pulmonary TB patient or inadequate treatment history with abnormal CXR). However, isoniazid prophylaxis will be not given based on positive TST or positive Quantiferon-Gold In-Tube assay.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or more
* Bone marrow transplant recipients

Exclusion Criteria:

* Recent contact of patients with active pulmonary tuberculosis
* Suspected active tuberculosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bone marrow transplant recipients
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
development of tuberculosis | after transplantation

SECONDARY OUTCOMES:
all cause mortality | after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee YM, Lee SO, Choi SH, Kim YS, Woo JH, Kim DY, Lee JH, Lee JH, Lee KH, Kim SH. A prospective longitudinal study evaluating the usefulness of the interferon-gamma releasing assay for predicting active tuberculosis in allogeneic hematopoietic stem cell transplant recipients. J Infect. 2014 Aug;69(2):165-73. doi: 10.1016/j.jinf.2014.02.019. Epub 2014 Mar 16. PMID 24647146
- [Derived] Moon SM, Lee SO, Choi SH, Kim YS, Woo JH, Yoon DH, Suh C, Kim DY, Lee JH, Lee JH, Lee KH, Kim SH. Comparison of the QuantiFERON-TB Gold In-Tube test with the tuberculin skin test for detecting latent tuberculosis infection prior to hematopoietic stem cell transplantation. Transpl Infect Dis. 2013 Feb;15(1):104-9. doi: 10.1111/j.1399-3062.2012.00765.x. Epub 2012 Jul 23. PMID 22823749